CLINICAL TRIAL: NCT00150579
Title: A Phase III, Randomized, Double-blind, Multi-center, Placebo-Controlled, Parallel-Group, Safety and Efficacy Study of SPD465 in Adults With Attention-Deficit Hyperactivity Disorder (ADHD).
Brief Title: Efficacy and Safety of SPD465 in Adults With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SPD465-301
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Amphetamine; Fumigant 93

INTERVENTIONS:
Drug: Neutral salts of dextroamphetamine sulfate, USP, amphetamine sulfate, USP, d-amphetamine saccharate, d, l-amphetamine aspartate monohydrate

SUMMARY:
The purpose of this study is to assess the safety and effectiveness of SPD465 compared to placebo (a capsule with no medication in it) in the treatment of ADHD. The study will also look at how SPD465 affects sleep and how the participants perceive their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of ADHD
* Baseline ADHD-RS-IV score >= 24
* Non-pregnant females of childbearing potential must comply with contraceptive restrictions

Exclusion Criteria:

* Significantly underweight or morbidly obese
* Comorbid psychiatric diagnosis with significant symptoms such as Axis II disorders or severe Axis I disorders
* History of seizure, tic disorder, or a current diagnosis and/or family history of Tourette's Disorder

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240
Dates: Start 2005-01-27 (Actual); Primary Completion 2005-06-14 (Actual); Study Completion 2005-06-14 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the ADHD-rating scale 4th Edition (ADHD-RS-IV) total score to the Endpoint assessment. | Baseline, and the Endpoint (average of weeks 5, 6, 7).
  The Endpoint is the average of the values obtained at Weeks 5, 6, and 7.

SECONDARY OUTCOMES:
Change from Baseline in the Clinical Global Impression of Improvement scale (CGI-I) to the Endpoint assessment. | Baseline, and the Endpoint (average of weeks 5, 6, 7).
  The Endpoint is the average of the values obtained at Weeks 5, 6, and 7.
Change from Baseline in the Time-Sensitive ADHD Symptom Scale (TASS) score to the Endpoint assessment. | Baseline, and the Endpoint (average of weeks 5, 6, 7).
  The Endpoint is the average of the values obtained at Weeks 5, 6, and 7.
Change from Baseline in the Brown Attention Deficit Disorder Scale (BADDS) to the Endpoint assessment | Baseline, and the Endpoint (average of weeks 5, 6, 7).
  The Endpoint is the average of the values obtained at Weeks 5, 6, and 7.
Change in Baseline in the Adult ADHD Impact Module (AIM-A) score to the Endpoint assessment | Baseline, and the Endpoint (average of weeks 5, 6, 7).
  The Endpoint is the average of the values obtained at Weeks 5, 6, and 7.
Change from Baseline in Pittsburgh Sleep Quality Index (PSQI) at Week 1 | Baseline and Week 1.
Change from Baseline in Pittsburgh Sleep Quality Index (PSQI) at Week 4 | Baseline and Week 4.
Change from Baseline in Pittsburgh Sleep Quality Index (PSQI) at Week 7 | Baseline and Week 7.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

REFERENCES:
- [Derived] Surman CBH, Robertson B, Chen J, Cortese S. Post-Hoc Analyses of the Effects of Baseline Sleep Quality on SHP465 Mixed Amphetamine Salts Extended-Release Treatment Response in Adults with Attention-Deficit/Hyperactivity Disorder. CNS Drugs. 2019 Jul;33(7):695-706. doi: 10.1007/s40263-019-00645-z. PMID 31228031
- [Derived] Brown TE, Landgraf JM. Improvements in executive function correlate with enhanced performance and functioning and health-related quality of life: evidence from 2 large, double-blind, randomized, placebo-controlled trials in ADHD. Postgrad Med. 2010 Sep;122(5):42-51. doi: 10.3810/pgm.2010.09.2200. PMID 20861587
- [Derived] Spencer TJ, Landgraf JM, Adler LA, Weisler RH, Anderson CS, Youcha SH. Attention-deficit/hyperactivity disorder-specific quality of life with triple-bead mixed amphetamine salts (SPD465) in adults: results of a randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2008 Nov;69(11):1766-75. doi: 10.4088/jcp.v69n1112. Epub 2008 Nov 4. PMID 19026251
- [Derived] Spencer TJ, Adler LA, Weisler RH, Youcha SH. Triple-bead mixed amphetamine salts (SPD465), a novel, enhanced extended-release amphetamine formulation for the treatment of adults with ADHD: a randomized, double-blind, multicenter, placebo-controlled study. J Clin Psychiatry. 2008 Sep;69(9):1437-48. doi: 10.4088/jcp.v69n0911. Epub 2008 Sep 9. PMID 19012813